CLINICAL TRIAL: NCT05670548
Title: Early Prediction of Postpartum Glucose Metabolism Abnormalities in Gestational Diabetes Mellitus Based on Gestational Metabolic Profile and Lipid Profile
Brief Title: Early Prediction of Postpartum Glucose Metabolism Abnormalities in Gestational Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-20220336-R
Record Dates: First submitted 2023-01-01; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, placenta, umbilical cord blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Abnormal postpartum glucose metabolism: GDM with positive OGTT results at 6-12 weeks postpartum
  Interventions: Other: Questionnaire survey and specimen collection
- Control: GDM with negative OGTT results at 6-12 weeks postpartum
  Interventions: Other: Questionnaire survey and specimen collection

INTERVENTIONS:
Other: Questionnaire survey and specimen collection — A questionnaire survey was conducted when pregnant women were enrolled, and blood were collected at 24-28 gestational weeks. Placenta and umbilical cord blood are collected during delivery.

SUMMARY:
This project is expected to screen reliable serum markers in pregnant women with gestational diabetes mellitus (GDM) by using metabolic profiling and lipid profiling clinical high-throughput mass spectrometry technology. We intend to build an early pregnancy prediction model for postpartum glucose metabolism abnormalities of GDM. At the same time, this project plans to develop a predictive management system based on this model, so that it can be widely used in clinical detection process, realize the advance of the early warning window period of abnormal glucose metabolism, and provide theoretical guidance for the early postpartum blocking of GDM to the outcome of abnormal glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Plan to have routine prenatal examinations and give birth in the research center
* GDM was diagnosed at 24-28 gestational weeks
* Singleton pregnancy
* Without other pregnancy complications
* Willing to cooperate with the hospital to follow up

Exclusion Criteria:

* Have diseases that affect metabolic function or even threaten the life of the mother and fetus before pregnancy, such as diabetes, heart disease, liver and kidney diseases, thyroid diseases with drug, autoimmune diseases, malignant tumors, AIDS, etc.
* Fetus has a known deformity or genetic defects
* Incomplete clinical data

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This project intends to recruit pregnant women with GDM who go to the research center for routine prenatal examination and OGTT screening at 24-28 gestational weeks.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum lipidomics | During the 24-28 geatational weeks.
  The differential serum lipid molecules in serum were detected by the self-developed detection chip, and the markers related to postpartum glucose metabolism abnormalities in GDM were screened. Specimens were collected during the 24-28 geatational weeks.
Serum metabolomics | During the 24-28 geatational weeks.
  The differential serum metabolism molecules in serum were detected by the self-developed detection chip, and the markers related to postpartum glucose metabolism abnormalities in GDM were screened. Specimens were collected during the 24-28 geatational weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoxia Liang, Prof., Study Director — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's Hospital School Of Medicine Zhejiang University, Hangzhou, Zhejiang, China